CLINICAL TRIAL: NCT03269591
Title: Electromagnetic Field Versus Diclofenac Drugs on Primary Dysmenorrhea: Arandomized Controlled Trial in the Egyptian Women
Brief Title: Electromagnetic Field Versus Diclofenac Drugs on Primary Dysmenorrhea
Acronym: magnetic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ghada Ebrahim El Refaye, Clinical lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: dr ghada
Record Dates: First submitted 2017-08-30; First posted 2017-09-01 (Actual); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Electromagnetic Field; Dysmenorrhea
Keywords: Dysmenorrhea; Pulsed electromagnetic field; Diclofenac
MeSH Terms: conditions — Dysmenorrhea | interventions — Diclofenac; Pain Measurement

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: (Participant, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Pulsed electromagnetic field (Active Comparator): magnetic therapy device which generate frequency from 5-100 Hz and intensity from 1 to 60 Gauss. Group (A) received 20 min 3 times per week for three month with strength 60 gauss and frequency 50 Hz
  Interventions: Device: Pulsed electromagnetic field; Drug: diclofenac tablets; Diagnostic Test: Visual analogue scale; Diagnostic Test: Progesterone blood level; Diagnostic Test: Menstrual symptom questionnaire
- diclofenac tablets (Experimental): (50 mg) few hours at the onset of menstruation for 3 months
  Interventions: Device: Pulsed electromagnetic field; Drug: diclofenac tablets; Diagnostic Test: Visual analogue scale; Diagnostic Test: Progesterone blood level; Diagnostic Test: Menstrual symptom questionnaire
- Visual analogue scale (Other): was used to determine the pain intensity level. Pain assessed before and after treatment procedure (3 month)
  Interventions: Device: Pulsed electromagnetic field; Drug: diclofenac tablets; Diagnostic Test: Visual analogue scale; Diagnostic Test: Progesterone blood level; Diagnostic Test: Menstrual symptom questionnaire
- Progesterone blood level (Other): Sample of blood was taken to detect the level of progesterone.
  Interventions: Device: Pulsed electromagnetic field; Drug: diclofenac tablets; Diagnostic Test: Visual analogue scale; Diagnostic Test: Progesterone blood level; Diagnostic Test: Menstrual symptom questionnaire
- Menstrual symptom questionnaire (Other): to assess symptoms of dysmenorrhea.
  Interventions: Device: Pulsed electromagnetic field; Drug: diclofenac tablets; Diagnostic Test: Visual analogue scale; Diagnostic Test: Progesterone blood level; Diagnostic Test: Menstrual symptom questionnaire

INTERVENTIONS:
Device: Pulsed electromagnetic field — EASY Qs portable (by ASA, Italy)
Drug: diclofenac tablets — drugs
Diagnostic Test: Visual analogue scale — a graphic rating scale
Diagnostic Test: Progesterone blood level — blood test
Diagnostic Test: Menstrual symptom questionnaire — questionnaire

SUMMARY:
Electromagnetic field versus diclofenac drugs on primary dysmenorrhea: Arandomized controlled trial in the Egyptian women

DETAILED DESCRIPTION:
Background: Primary dysmenorrhea is one of the most common complaints of women and is also the most common gynecological problem worldwide. These cramps are recurrent and 90% adolescent girls and about 50% women suffer from it. Purpose of the study: to determine which is more effective in alleviating primary dysmenorrhea; pulsed electromagnetic field or diclofenac drugs. Methodology: The study was a randomized, double-blinded trial, fifty adult females participated in this study, were divided randomly into two groups equal in numbers: group (A) received pulsed electromagnetic field applied on pelvic region, 3 times per week for 3 months, 20 minutes per day and group (B) received diclofenac tablets, 50 mg only with onset of menstrual pain. All participants in both groups (A and B) were assessed pre- and post-treatment through measuring progesterone level in the blood, assessment of pain using visual analogue scale and physical as well as psychological symptoms by using menstrual symptom questionnaire.

ELIGIBILITY:
Inclusion Criteria:

-regular menstrual cycle 21-35 days lasting 3-7 days

Exclusion Criteria:

* Irregulars or infrequent menstrual cycles, Pacemaker, Myasthenia gravis, hyperthyroidism, active tuberculosis and psychosis

Ages: 17 Years to 24 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — females
Enrollment: 50 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-10-29 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale | three months
  was used to determine the pain intensity level. Pain assessed before and after treatment procedure (3 month); in both groups (A and B) by (16), it is a graphic rating scale with numerical values placed equidistantly along the line. The descriptors and numbers help the subject to place her estimate on line in which (0) mean no pain, (1) equal mild pain, (2) equal moderate pain, (3) mean severe pain and (4) mean unbearable pain.

SECONDARY OUTCOMES:
Progesterone blood level | three months
  Sample of blood was taken to detect the level of progesterone.
Menstrual symptom questionnaire | three months
  to assess symptoms of dysmenorrhea

IPD SHARING:
Plan to Share IPD: Yes
Electromagnetic field versus diclofenac drugs on primary dysmenorrhea: Arandomized controlled trial in the Egyptian women
Supporting Information: Study Protocol
Time Frame: three months
Access Criteria: the protocol of study, for 3 months